CLINICAL TRIAL: NCT04655027
Title: ALTAI: An Open-Label, Randomized, Active-Controlled, Parallel Design, Multicenter Phase IV Study to Investigate the Effect of Roxadustat Versus Recombinant Human Erythropoietin (rHuEPO) on Oral Iron Absorption in Chinese Patients With Anemia of Chronic Kidney Disease (CKD)
Brief Title: A Study to Investigate the Effect of Roxadustat Versus Recombinant Human Erythropoietin (rHuEPO) on Oral Iron Absorption in Chinese Patients With Anemia of Chronic Kidney Disease (CKD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5741C00002
Record Dates: First submitted 2020-12-03; First posted 2020-12-04 (Actual); Results first posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Anemia of Chronic Kidney Disease
Keywords: Recombinant Human Erythropoietin; Roxadustat; Coronavirus disease of 2019; Chronic kidney disease; Anemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia | interventions — roxadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Roxadustat (Experimental): Patients will receive oral dose of roxadustat three times a week (TIW) for 2- weeks during treatment period.
  Interventions: Drug: Roxadustat
- rHuEPO (Active Comparator): Patients will receive uniform brand of short acting intravenous or subcutaneous dose of rHuEPO two times a week (BIW) or TIW based upon their previous dose of rHuEPO for 2- weeks during treatment period.
  Interventions: Drug: rHuEPO

INTERVENTIONS:
Drug: Roxadustat — The starting dose of roxadustat will be in accordance with the China package insert, and will depend on the body weight of the patient: 100 mg (45 to < 60 kg) or 120 mg (≥ 60 kg) in patients on dialysis; 70 mg (40 to < 60 kg) or 100 mg (≥ 60 kg) in non-dialysis patients.
  Arms: Roxadustat
Drug: rHuEPO — The starting dose of rHuEPO will be in accordance to the dosage approved in rHuEPO China package insert (patients on weekly dose of 6000 IU [dosing will BIW], and patients on weekly dose of >6000 IU [dosing will TIW]) and on patient's haemoglobin levels.
  Arms: rHuEPO

SUMMARY:
This is a Phase IV, randomized, active-controlled, open-label, parallel design, multicenter prospective study to evaluate the effect of roxadustat versus rHuEPO treatment on the gastrointestinal (GI) iron absorption in patients with anemia of Stage 4 and Stage 5 CKD.

DETAILED DESCRIPTION:
This is an open-label study, after eligibility confirmation patients will be randomized in a 1:1 ratio to either roxadustat or rHuEPO arms for 2 weeks.

The study will enroll eligible dialysis and non-dialysis patients ≥18 years of age, who have anemia of CKD, and are either dialysis-dependent (DD) and on a stable dose of rHuEPO within 4 weeks prior to screening, or are non-dialysis-dependent (NDD) and are being treated with rHuEPO (ie, on a stable dose of rHuEPO within 4 weeks prior to screening), or are rHuEPO -naïve at the time of screening.

Each patient will be contacted before the first Screening Visit (Visit 1) for the symptoms of coronavirus disease of 2019 (COVID-19) and for any contact with COVID-19 positive person within the past 14 days.

For each patient, the duration of participation in the study will be approximately 8 to 9 weeks divided into 3 periods: Screening Period (approximately 2-3 weeks); Treatment Period (2 weeks) and Post-Treatment Follow-up Period (4 weeks).

ELIGIBILITY:
Inclusion Criteria:

Informed consent • Provision of signed and dated, written informed consent form (ICF) prior to any mandatory study specific procedures, sampling, and analyses.

Type of patient and disease characteristics

At Visit 1 prior to screening

Dialysis patients:

* Patients receiving hemodialysis (HD) or peritoneal dialysis (PD) for treatment of end-stage renal disease (ESRD) for at least 12 weeks. Patients treated with HD must have access consisting of an arteriovenous (AV) fistula, AV graft, or tunneled (permanent) catheter. Patients on PD must have a functioning PD catheter in place.
* Hemodialysis patients should be on 3x/week dialysis with evidence of achievement of adequate dialysis as defined by standardized Kt/V ≥2.1 in HD, and total (renal + PD) weekly Kt/V ≥1.7 in PD documented twice during the 16 weeks preceding screening for the study.
* Patients should be on a stable rHuEPO dose as defined by change in rHuEPO dose, not exceeding 20% within 4 weeks prior to screening.

Non-dialysis patients:

* Patients with estimated glomerular filtration rate (eGFR) <30 mL/minute/1.73 m^2, corresponding to Stage 4 or Stage 5 CKD according to the Kidney Disease Outcomes Quality Initiative (KDOQI), and not receiving dialysis.
* Patients should either be on a stable dose of rHuEPO for 4 weeks before screening or be rHuEPO-naïve.

Dialysis and non-dialysis patients:

• Patients agree not to take any new traditional Chinese medicine (TCM) and not to change, dose, schedule or brand of any TCM from beginning of the Screening Period through the end of the Follow-up Period.

At Visit 1 (screening)

* Ferritin ≥50 ng/mL and transferrin saturation (TSAT) ≥15% in non-dialysis patients
* Ferritin ≥100 ng/mL and TSAT ≥20% in dialysis patients.
* Dry body weight should be 45 to 100 kg.

During the Screening Period:

* Dialysis patients must have a mean Hb level of ≥ 9 to ≤ 12 g/dL based on the mean of the 2 most recent central laboratory Hb values within 0.50 g/dL on 2 assays taken at least 7 days apart during the Screening Period.
* Non-dialysis patients must have a mean Hb level of ≥ 9 to ≤ 12 g/dL for rHuEPO-user patients and ≥ 7 and ≤ 10 g/dL for rHuEPO-naïve patients, based on the mean of the 2 most recent central laboratory Hb values within 0.50 g/dL on 2 assays taken at least 7 days apart during the Screening Period.

At Visit 1 Screening:

* Serum folate level ≥ lower limit of normal (LLN).
* Serum vitamin B12 level ≥ LLN.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 3 x ULN and total bilirubin (TBL) ≤ 1.5 x ULN.
* Negative test results on the swab test to rule out active COVID-19 infection. If according to site procedures the test for COVID-19 infection cannot be performed at the first Screening Visit, the test should be performed as soon as possible thereafter but must be performed before the patient returns for the next study visit. Any patient who has had confirmed COVID-19 infection in the past, has fully recovered from symptoms at least 14 days prior to Screening, and has a negative swab test result for COVID-19 infection at Screening, may be included in the study.

Reproduction:

* Serum pregnancy test should be negative for female of childbearing potential at the start of the Screening Period.
* Female patients of childbearing potential and male patients (non-surgically sterile) with a female partner of childbearing potential must, if not practicing complete sexual abstinence, agree to practice a dual method of contraception.

Contraceptive methods must be practiced upon being randomized to the study and through 7 days after the last dose of study treatment. Male patients must not donate or bank sperm during this same time period.

Exclusion Criteria:

Medical conditions

* New York Heart Association Class III or IV congestive heart failure (CHF) at screening.
* Acute coronary syndrome, stroke, seizure or a thrombotic/thromboembolic event (eg, deep vein thrombosis or pulmonary embolism) within 12 weeks prior to randomization.
* History of severe, chronic, end-stage, or uncontrolled autoimmune liver disease with ALT 3 x ULN, or AST > 3 × ULN, or total bilirubin > 1.5 × ULN.
* Known hereditary hematologic disease such as thalassemia, sickle cell anemia, a history of pure red-cell aplasia or other known causes for anemia other than CKD.
* Known and untreated retinal vein occlusion or known and untreated proliferative diabetic retinopathy.
* Systolic BP ≥160 mmHg or diastolic BP ≥95 mmHg (confirmed by repeated measurement), within 2 weeks prior to randomization. Patients may be rescreened once BP is controlled.
* History of prostate cancer, breast cancer, renal cell carcinoma or any other malignancy, except the following: cancers determined to be cured or in remission for ≥5 years; curatively resected basal cell or squamous cell skin cancers, cervical cancer in situ, or resected colonic polyps.
* Chronic inflammatory diseases such as rheumatoid arthritis, systemic lupus erythromatosus (SLE), ankylosing spondylitis, psoriatic arthritis or active inflammatory bowel disease that is determined to be the principal cause of anemia.
* Known hemosiderosis, hemochromatosis or hypercoagulable condition.
* Any prior organ transplant or a scheduled organ transplantation date.
* Any current condition leading to active significant blood loss.
* Known allergy to the study treatment or any of its ingredients.
* Any medical condition, including active, clinically significant infection, that in the opinion of the Investigator or Sponsor may pose a safety risk to a patient in this study, which may confound safety or efficacy assessment or may interfere with study participation.
* Intolerance of oral iron in the past as defined by stomach upset, nausea, vomiting, or diarrhea.
* Active GI bleed.
* Hospitalizations within the 12 weeks preceding study randomization for GI bleeding or Congestive heart failure.
* Life expectancy <6 months.
* Patients who are likely to be initiated on dialysis within the next 3 months per Investigator's assessment at the time of screening.
* Previous bowel resection.
* Coeliac disease.
* Gastroenteritis in the 4 weeks prior to randomization.
* Cognitive disabilities, physical or psychiatric disease that in the opinion of the Investigator/clinician influence the patient's adherence and successful completion of the study.

Prior/concomitant therapy:

* Any treatment with roxadustat or a Hypoxia-Inducible Factor Prolyl Hydroxylase Inhibitors (HIF-PHI).
* Any red blood cells transfusion within 6 weeks prior to the first Screening Visit, or during the Screening Period.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within the 12 weeks prior to Screening Visit.
* Exposure to IV iron or use of TRIFERIC® in dialysate during the Screening Period (ie, 2 weeks before randomization [Day 1]).
* Exposure to iron-chelating agent (eg, deferoxamine/desferrioxamine, deferiprone or deferaxirox therapy) within the 6 weeks prior to the first Screening Visit.

Prior/concurrent clinical study experience:

• Participation in any other clinical study that included drug treatment within at least 4 weeks of screening.

Other exclusions:

* Involvement in the planning and/or conduct of the study (applies to AstraZeneca and FibroGen staff and/or staff at the study site).
* Patient non-adherence to medications or missing >1 dialysis treatments/month per the Investigator's knowledge.
* Previous randomization in the present study.
* History of alcohol or drug abuse within 2 years prior to randomization.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li Xuemei, Principal Investigator — Peking Union Medical College Hospital (Dongdan campus) No.1 Shuaifuyuan Wangfujing Dongcheng District Beijing, China 100730
Locations (6):
- China (6):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Guangzhou
  - Research Site, Jinan
  - Research Site, Shenyang
  - Research Site, Wuhan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Wu H, Cheng H, Wang C, Yao L, Qin S, Zuo L, Hu Z, Zhang C, Wu Y, Hofherr A, Mohan K, Rush S, Li X. Roxadustat and Oral Iron Absorption in Chinese Patients with Anemia of Chronic Kidney Disease: A Randomized, Open-Label, Phase 4 Study (ALTAI). Adv Ther. 2024 Mar;41(3):1168-1183. doi: 10.1007/s12325-023-02741-5. Epub 2024 Jan 27. PMID 38280066
- See also: redacted Statistical Analysis Plan — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5741C00002&attachmentIdentifier=2a566fb7-52ad-41c2-812d-7d85e0e91770&fileName=redacted_Statistical_Analysis_Plan.pdf&versionIdentifier=
- See also: redacted Clinical Study Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5741C00002&attachmentIdentifier=a2c390ba-c2c0-494d-a275-108c75d90b55&fileName=redacted_Clinical_Study_Protocol.pdf&versionIdentifier=
- See also: redacted Clinical Study Report Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5741C00002&attachmentIdentifier=bda09028-f356-4e0f-a2d8-71d619a2b68f&fileName=redacted_Clinical_Study_Report_Synopsis.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 25 subjects at 8 clinical sites in China, of which 5 sites enrolled patients from 17 March 2021 (first subject first randomized) to 12 October 2021 (last subject last visit).
Pre-assignment Details: The screening period was up to 3 weeks. All the study assessments were performed as per the schedule of assessment. Eligible patients were randomized at a 1:1 ratio to receive either Roxadustat or rHuEPO [Recombinant Human Erythropoietin] for 14 days starting from Day 1.
Groups:
- Roxadustat: Patients received oral dose of Roxadustat tablets three times a week (TIW) for 2 weeks during treatment period and followed 4 weeks of follow up period.
- rHuEPO: Patients received uniform brand of short acting intravenous or subcutaneous dose of rHuEPO two times a week (BIW) or TIW based upon their previous dose of rHuEPO for 2 weeks during treatment period and followed 4 weeks of follow up period.
Period: Overall Study
Arm/Group | Roxadustat | rHuEPO
Started | 13 | 12
Completed | 12 | 12
Not Completed | 1 | 0
Not completed — Failure to meet inclusion/exclusion criteria/ Due to COVID-19 pandemic | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Full analysis Set (FAS) was the primary efficacy analysis set and included all randomized patients who completed baseline (Day 1) measurements for any efficacy analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Roxadustat | rHuEPO | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.3 (12.09) | 52.8 (12.64) | 55.1 (12.32)
Age, Customized [Count of Participants; unit: Participants]
  ≥ 18 to < 50 years | 5 | 4 | 9
  ≥ 50 to < 65 years | 3 | 6 | 9
  ≥ 65 to < 75 years | 4 | 2 | 6
  ≥ 75 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 4 | 5 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Difference From Baseline to Day 15 in Area Under Curve (AUC) of GI Iron Absorption (0-3 Hours)
Description: The main effect of roxadustat versus rHuEPO on GI iron absorption was evaluated.
Time Frame: From Baseline (Day 1) to Day 15
Population: The FAS was the primary efficacy analysis set and included all randomized patients who completed baseline (Day 1) measurements for any efficacy analysis.
  Here, the number analyzed signified only the subjects with available data that were evaluated on that specific group.
Measure: Mean (Standard Deviation); unit: gram*3hours/deciliter (g*3hr/dL)
Arm/Group | Roxadustat | rHuEPO
Number analyzed (Participants) | 12 | 11
gram*3hours/deciliter (g*3hr/dL)
  Change from baseline | 11.288 (28.1506) | -0.259 (9.7369)
  Hemodialysis (HD) group- Change from baseline: number analyzed (Participants) | 4 | 6
  Hemodialysis (HD) group- Change from baseline | 20.125 (29.9536) | -1.625 (10.2189)
  Peritoneal dialysis (PD)- Change from baseline: number analyzed (Participants) | 6 | 4
  Peritoneal dialysis (PD)- Change from baseline | -2.408 (19.4973) | -2.263 (6.7321)
  Non-dialysis-dependent (NDD)- Change from baseline: number analyzed (Participants) | 2 | 1
  Non-dialysis-dependent (NDD)- Change from baseline | 34.700 (39.8808) | 15.950 (NA) — As only 1 participant was evaluable, hence SD was not calculable.
Statistical Analysis 1: Comparison: Roxadustat vs rHuEPO; Test type: Other — Treatment effect; p = 0.212, ANCOVA; Difference in Estimate (LSM) = 19.50, 95% CI 2-sided [-11.155 to 50.150], Standard Error of Mean 15.62

2. Secondary Outcome: Difference From Baseline to Day 15 in Area Under Curve (AUC) of Iron Absorption (0-3 Hours)
Description: The effect and interaction with key baseline variables of roxadustat versus rHuEPO on iron absorption was assessed.
Time Frame: From Baseline (Day 1) to Day 15
Population: The FAS was the primary efficacy analysis set and included all randomized patients who completed baseline (Day 1) measurements for any efficacy analysis.
  Here, the number analyzed signified only the subjects with available data that were evaluated for this specific outcome measure.
  The change from baseline reported uses observed values only, which is only defined when both Baseline and Day 15 values are non-missing.
Measure: Mean (Standard Deviation); unit: gram*3hours/deciliter (g*3hr/dL)
Arm/Group | Roxadustat | rHuEPO
Number analyzed (Participants) | 12 | 11
gram*3hours/deciliter (g*3hr/dL) | 11.288 (28.1506) | -0.259 (9.7369)
Statistical Analysis 1: Comparison: Roxadustat vs rHuEPO; Test type: Other — Baseline hepcidin by treatment effect; p = 0.441, ANCOVA; Difference in Estimate = -0.13, 95% CI 2-sided [-0.477 to 0.208], Standard Error of Mean 0.17
Statistical Analysis 2: Comparison: Roxadustat vs rHuEPO; Test type: Other — Baseline hs CRP by treatment effect; p = 0.532, ANCOVA; Difference in Estimates = -2.34, 95% CI 2-sided [-9.707 to 5.017], Standard Error of Mean 3.76

3. Secondary Outcome: Difference From Baseline to Day 15 in Serum Iron
Description: The effect and interaction with baseline variables of roxadustat versus rHuEPO on the indices of iron metabolism: serum iron was assessed.
Time Frame: From baseline (Day 1) to Day 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micromole/Liter (µmol/L)
Arm/Group | Roxadustat | rHuEPO
Number analyzed (Participants) | 13 | 11
micromole/Liter (µmol/L) | 2.077 (7.9263) | -0.845 (7.6225)
Statistical Analysis 1: Comparison: Roxadustat vs rHuEPO; Test type: Other — Treatment effect; p = 0.688, Geometric ANCOVA; Geometric ANCOVA of relative change from baseline. The Standard error of Mean (SEM) refers to Geometric SEM; Ratio of Estimates = 1.09, 95% CI 2-sided [0.723 to 1.635], Standard Error of Mean 1.23
Statistical Analysis 2: Comparison: Roxadustat vs rHuEPO; Test type: Other — Baseline hepcidin-by-treatment effect; p = 0.029, ANCOVA; Difference in Estimates = 0.43, 95% CI 2-sided [0.045 to 0.822], Standard Error of Mean 0.20
Statistical Analysis 3: Comparison: Roxadustat vs rHuEPO; Test type: Other — Baseline hs-CRP-by-treatment effect; p = 0.568, ANCOVA; Difference in Estimates = 0.08, 95% CI 2-sided [-0.201 to 0.366], Standard Error of Mean 0.14

4. Secondary Outcome: Difference From Baseline to Day 15 in Ferritin
Description: The effect and interaction with baseline variables of roxadustat versus rHuEPO on the indices of iron metabolism: Ferritin was assessed.
Time Frame: From baseline (Day 1) to Day 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: microgram/Liter (µg/L)
Arm/Group | Roxadustat | rHuEPO
Number analyzed (Participants) | 13 | 11
microgram/Liter (µg/L) | -49.354 (175.3039) | -43.536 (79.3449)
Statistical Analysis 1: Comparison: Roxadustat vs rHuEPO; Test type: Other — Treatment effect; p = 0.096, Geometric ANCOVA; Geometric ANCOVA of relative change from baseline. The Standard error of Mean (SEM) refers to Geometric SEM; Ratio of Estimates = 0.84, 95% CI 2-sided [0.687 to 1.031], Standard Error of Mean 1.11
Statistical Analysis 2: Comparison: Roxadustat vs rHuEPO; Test type: Other — Baseline hepcidin-by-treatment effect; p = 0.630, ANCOVA; Difference in Estimates = -0.06, 95% CI 2-sided [-0.282 to 0.171], Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: Roxadustat vs rHuEPO; Test type: Other — Baseline hs-CRP-by-treatment effect; p = 0.015, ANCOVA; Difference in Estimates = 0.19, 95% CI 2-sided [0.037 to 0.342], Standard Error of Mean 0.08

5. Secondary Outcome: Difference From Baseline to Day 15 in Total Iron Binding Capacity (TIBC)
Description: The effect and interaction with baseline variables of roxadustat versus rHuEPO on the indices of iron metabolism: TIBC was assessed.
Time Frame: From baseline (Day 1) to Day 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micromole/Liter (µmol/L)
Arm/Group | Roxadustat | rHuEPO
Number analyzed (Participants) | 13 | 10
micromole/Liter (µmol/L) | 8.638 (5.1118) | -0.490 (3.7784)
Statistical Analysis 1: Comparison: Roxadustat vs rHuEPO; Test type: Other — Treatment effect; p < 0.001, Geometric ANCOVA; Geometric ANCOVA of relative change from baseline. The Standard error of Mean (SEM) refers to Geometric SEM; Ratio of Estimates = 1.23, 95% CI 2-sided [1.123 to 1.354], Standard Error of Mean 1.05
Statistical Analysis 2: Comparison: Roxadustat vs rHuEPO; Test type: Other — Baseline hepcidin-by-treatment effect; p = 0.171, ANCOVA; Difference in Estimates = 0.06, 95% CI 2-sided [-0.027 to 0.149], Standard Error of Mean 0.04
Statistical Analysis 3: Comparison: Roxadustat vs rHuEPO; Test type: Other — Baseline hs-CRP-by-treatment effect; p = 0.387, ANCOVA; Difference in Estimates = 0.03, 95% CI 2-sided [-0.039 to 0.101], Standard Error of Mean 0.04

6. Secondary Outcome: Relative Difference From Baseline to Day 15 in Transferrin Saturation (TSAT)
Description: The effect and interaction with baseline variables of roxadustat versus rHuEPO on the indices of iron metabolism: TSAT (fraction of TIBC) was assessed.
Time Frame: From baseline (Day 1) to Day 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Roxadustat | rHuEPO
Number analyzed (Participants) | 13 | 10
Ratio | -0.024 (0.1806) | -0.030 (0.2007)
Statistical Analysis 1: Comparison: Roxadustat vs rHuEPO; Test type: Other — Treatment effect; p = 0.561, Geometric ANCOVA; Geometric ANCOVA of relative change from baseline. The Standard error of Mean (SEM) refers to Geometric SEM; Ratio of Estimates = 0.89, 95% CI 2-sided [0.606 to 1.312], Standard Error of Mean 1.22
Statistical Analysis 2: Comparison: Roxadustat vs rHuEPO; Test type: Other — Baseline hepcidin-by-treatment effect; p = 0.043, ANCOVA; Difference in Estimates = 0.38, 95% CI 2-sided [0.013 to 0.750], Standard Error of Mean 0.19
Statistical Analysis 3: Comparison: Roxadustat vs rHuEPO; Test type: Other — Baseline hs-CRP-by-treatment effect; p = 0.766, ANCOVA; Difference in Estimates = 0.04, 95% CI 2-sided [-0.222 to 0.302], Standard Error of Mean 0.13

7. Secondary Outcome: Difference From Baseline to Day 15 in Transferrin
Description: The effect and interaction with baseline variables of roxadustat versus rHuEPO on the indices of iron metabolism: Transferrin was assessed.
Time Frame: From baseline (Day 1) to Day 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: gram/Liter (g/L)
Arm/Group | Roxadustat | rHuEPO
Number analyzed (Participants) | 13 | 12
gram/Liter (g/L) | 0.452 (0.3550) | -0.012 (0.1393)
Statistical Analysis 1: Comparison: Roxadustat vs rHuEPO; Test type: Other — Treatment effect; p < 0.001, Geometric ANCOVA; Geometric ANCOVA of relative change from baseline. The Standard error of Mean (SEM) refers to Geometric SEM; Ratio of Estimates = 1.23, 95% CI 2-sided [1.108 to 1.369], Standard Error of Mean 1.05
Statistical Analysis 2: Comparison: Roxadustat vs rHuEPO; Test type: Other — Baseline hepcidin-by-treatment effect; p = 0.351, ANCOVA; Difference in Estimates = 0.05, 95% CI 2-sided [-0.059 to 0.159], Standard Error of Mean 0.05
Statistical Analysis 3: Comparison: Roxadustat vs rHuEPO; Test type: Other — Baseline hs-CRP-by-treatment effect; p = 0.248, ANCOVA; Difference in Estimates = 0.04, 95% CI 2-sided [-0.031 to 0.114], Standard Error of Mean 0.03

8. Secondary Outcome: Difference From Baseline to Day 15 in Soluble Transferrin Receptor
Description: The effect and interaction with baseline variables of roxadustat versus rHuEPO on the indices of iron metabolism: Soluble transferrin receptor was assessed.
Time Frame: From baseline (Day 1) to Day 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligram/Liter (mg/L)
Arm/Group | Roxadustat | rHuEPO
Number analyzed (Participants) | 13 | 12
milligram/Liter (mg/L) | 1.876 (3.0627) | 0.466 (0.5556)
Statistical Analysis 1: Comparison: Roxadustat vs rHuEPO; Test type: Other — Treatment effect; p = 0.021, Geometric ANCOVA; Geometric ANCOVA of relative change from baseline. The Standard error of Mean (SEM) refers to Geometric SEM; Ratio of Estimates = 1.29, 95% CI 2-sided [1.043 to 1.598], Standard Error of Mean 1.11
Statistical Analysis 2: Comparison: Roxadustat vs rHuEPO; Test type: Other — Baseline hepcidin-by-treatment effect; p = 0.826, ANCOVA; Difference in Estimates = -0.03, 95% CI 2-sided [-0.276 to 0.223], Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: Roxadustat vs rHuEPO; Test type: Other — Baseline hs-CRP-by-treatment effect; p = 0.634, ANCOVA; Difference in Estimates = -0.04, 95% CI 2-sided [-0.212 to 0.132], Standard Error of Mean 0.08

9. Secondary Outcome: Difference From Baseline to Day 15 in Hepcidin
Description: The effect and interaction with baseline variables of roxadustat versus rHuEPO on the indices of Hepcidin was assessed.
Time Frame: From baseline (Day 1) to Day 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: microgram/Liter (µg/L)
Arm/Group | Roxadustat | rHuEPO
Number analyzed (Participants) | 13 | 12
microgram/Liter (µg/L) | -78.769 (87.9264) | -44.239 (88.2325)
Statistical Analysis 1: Comparison: Roxadustat vs rHuEPO; Test type: Other — Treatment effect; p = 0.007, Geometric ANCOVA; Geometric ANCOVA of relative change from baseline. The Standard error of Mean (SEM) refers to Geometric SEM; Ratio of Estimates = 0.45, 95% CI 2-sided [0.257 to 0.786], Standard Error of Mean 1.31
Statistical Analysis 2: Comparison: Roxadustat vs rHuEPO; Test type: Other — Baseline hepcidin-by-treatment effect; p = 0.610, ANCOVA; Difference in Estimates = -0.16, 95% CI 2-sided [-0.798 to 0.480], Standard Error of Mean 0.31
Statistical Analysis 3: Comparison: Roxadustat vs rHuEPO; Test type: Other — Baseline hs-CRP-by-treatment effect; p = 0.740, ANCOVA; Difference in Estimates = 0.07, 95% CI 2-sided [-0.387 to 0.536], Standard Error of Mean 0.22

10. Secondary Outcome: Number of Subjects With Adverse Events (AEs)
Description: AEs as variables of safety was assessed.
Time Frame: From screening (Starting on Day -21) until follow up (28 days) (approximately 7 weeks)
Population: The Safety analysis set included all randomized patients who received at least 1 dose of study treatment, with patients being analyzed as treated, rather than as randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Roxadustat | rHuEPO
Number analyzed (Participants) | 13 | 12
Participants
  Any AE | 5 | 2
  Any AE with outcome of death | 0 | 0
  Any Serious Adverse event (SAE) (including events with outcome of death) | 0 | 0
  Any AE leading to discontinuation of study treatment | 0 | 0
  Any AE leading to dose interruption | 0 | 0
  Any AE leading to dose reduction | 0 | 0
  Any AE leading to dose escalation | 0 | 0
  Any AE leading to withdrawal from study | 0 | 0
  Any AE possibly related to study treatment | 1 | 0

ADVERSE EVENTS:
Time Frame: From screening (Starting on Day -21) until follow up (28 days) (approximately 7 weeks)
Arm/Group | Roxadustat | rHuEPO
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 5/13 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Roxadustat (N=13) | rHuEPO (N=12)
Abdominal infection (Infections and infestations) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Open angle glaucoma (Eye disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
* NDD randomization strata were merged because recruitment was insufficient.
* The log-transform of AUC was removed from the primary assessment post-database-lock when negative AUC were discovered (which invalidated log-transformation).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This document contains trade secrets and confidential commercial information, disclosure of which is prohibited without providing advance notice to AstraZeneca and opportunity to object.

DOCUMENTS (2):
  • Study Protocol (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT04655027/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/27/NCT04655027/SAP_001.pdf